CLINICAL TRIAL: NCT06334601
Title: Diurnal Evaluation of Obstructive Sleep Apnea (OSA) Upper Airway Collapsibility and Muscle Responsiveness
Brief Title: Diurnal Evaluation of OSA Upper Airway Collapsibility and Muscle Responsiveness
Acronym: Muscle-OSA
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C333
Record Dates: First submitted 2024-03-19; First posted 2024-03-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Collapsibility of upper airways; Muscle responsiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive Sleep Apnea: Patients evaluated for sleep disorders, who present an at home-polygraphy with at least one EEG channel (PSG) reporting moderate-to severe obstructive sleep apnea (apnea-hypopnea index >14).
  Interventions: Diagnostic Test: Tests of upper airway collapsibility and muscle responsiveness.

INTERVENTIONS:
Diagnostic Test: Tests of upper airway collapsibility and muscle responsiveness. — Upper airway collapsibility, upper airway muscle responsiveness and loop gain will be assessed during single study visit.
  Polysomnography

SUMMARY:
In the framework of pathophysiological trait in obstructive sleep apnea (OSA) patients, a simplified method is proposed to measure upper airway (UA) collapsibility and muscle responsiveness during wakefulness.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep Apnea (OSA)
* At home-polygraphy with at least one EEG channel (PSG) reporting moderate-to severe obstructive sleep apnea (apnea-hypopnea index >14).

Exclusion Criteria:

* OSA treatment ongoing during two weeks before PSG
* Unstable cardio-respiratory disease in the 3 months before enrollment
* Subjects in O2 treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients evaluated for sleep disorders in our Institution, who present an at home-polygraphy with at least one EEG channel (PSG) reporting moderate-to severe obstructive sleep apnea (apnea-hypopnea index >14)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper airway collapsibility | During the diagnostic test
  Evaluation during wakefulness
Upper airway muscle responsiveness | During the diagnostic test
  Evaluation during wakefulness

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano,Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: No